CLINICAL TRIAL: NCT00184834
Title: Quality of Life After Surgical Treatment of Colorectal Liver Metastases
Brief Title: Quality of Life and Liver Metastases
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Other Study IDs: qol1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Colorectal Liver Metastases; Quality of Life
Keywords: colorectal; liver; metastases; health-related quality of life; surgery
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: quality of life

SUMMARY:
An increasing aggressiveness in the surgical approach of colorectal liver metastases is observed. This seems only justified when, besides prolongation of survival, also the health status of patients is considered. The aim of this prospective study is to investigate the impact of surgery on health-related quality of life in this specific patient population operated for colorectal liver metastases.Furthermore, as the indications for hepatic resection are broadened and patients with more extensive liver disease are operated on, the chance of non operable disease at laparotomy will increase. The effects of such an event on HRQol are also studied.

DETAILED DESCRIPTION:
In a prospective study several patients groups were identified. Patients undergoing liver resection and/or local ablative therapy. Patients with non operable disease at (explorative) laparotomy and outpatients with non operable disease as shown during work up for liver resection. Several validated instruments on HRQoL were ompleted preoperatively (baseline), a half month after operation and then every three months.

ELIGIBILITY:
Inclusion Criteria:

colorectal liver metastases (operable and non operable disease) and participation by means of filling in quality of life instruments

Exclusion Criteria:

drop out and therefore loss of quality of life instruments

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1999-06; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Langenhoff BS, Krabbe PF, Wobbes T, Ruers TJ. Quality of life as an outcome measure in surgical oncology. Br J Surg. 2001 May;88(5):643-52. doi: 10.1046/j.1365-2168.2001.01755.x. PMID 11350434